CLINICAL TRIAL: NCT06935201
Title: Get Back, A Digital Person-Centered Rehabilitation Program to Increase Physical Activity After Lumbar Spinal Stenosis Surgery - a Randomized Controlled Trial
Brief Title: Evaluation of a Digital Person-Centered Rehabilitation Program Targeting Physical Activity in Spinal Stenosis Surgery (Get Back)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sophiahemmet University (Other)
Collaborators: The Swedish Research Council (Other Government); University of Gothenburg Center for Person-Centred Care, GPCC (Unknown)
Responsible Party: Principal Investigator, Mari Lundberg, Professor, Sophiahemmet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Get Back RCT
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Spinal Stenosis Lumbar
Keywords: Rehabilitation; Person-centred care; Physical activity; Steps per day; Behavioral medicine; Telerehabilitation; Telehealth
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Get Back) (Experimental): The intervention includes up to 5 core sessions (video call) and 5 booster sessions (telephone) over 13 weeks (approx. 1 week before until 12 weeks after surgery). All sessions will be led by a physical therapist. The focus of each core session (1-5) is as follows:
  1. To establish the patient as an active, equal partner in the treatment and to formulate a shared health plan according to person-centered care.
  2. To follow up with postoperative analysis and activity initiation.
  3. To support graded physical activity by analysis, problem-solving, and behavioral strategies.
  4. To support graded physical activity by analysis, problem-solving, and behavioral strategies.
  5. To support the patient to independently continue with activity progress towards long term health and to formulate a maintenance plan.
  Interventions: Behavioral: Get Back
- Control (standard physical therapy) (No Intervention): The control group will follow standard physical therapy, meaning physical therapy as it is provided at each recruiting site when undergoing surgery due to spinal stenosis. As this may differ substantially between clinical sites nationally, data on frequency of physical therapy and the content of the physical therapy sessions during the study period will be collected as a control variable from the control group.

INTERVENTIONS:
Behavioral: Get Back — A rehabilitation program, targeting physical activity behavior, with a person-centered approach led by a physical therapist during 12 weeks (1 week before surgery until 12 weeks after surgery) in a digital format.
  Arms: Intervention (Get Back)

SUMMARY:
This study aims to investigate whether Get Back is more effective than standard rehabilitation in increasing the number of steps per day, improving physical activity levels, and functional ability for patients undergoing surgery for lumbar spinal stenosis (LSS). LSS is common, especially among older adults, leading to increased health risks and reduced quality of life. Despite its prevalence (about 60% of all spinal surgeries in Sweden), many LSS patients remain physically inactive post-surgery, worsening their health. Rehabilitation remains a global challenge with unequal access, and many patients feel disengaged from the process. Get Back is a digital rehabilitation program including three components: gradually increasing physical activity, managing fear and avoidance behaviors, and using behavior change techniques. It has shown promising results in a pilot study, increasing daily steps. The program uses a person-centered approach tailored to personal needs. This multicenter randomized controlled trial will assess efficacy, process, and cost-effectiveness. It will also explore how preoperative values such as physical capacity and psychological factors predict changes in daily steps after surgery. Data will be collected via questionnaires, functional tests, and interviews, with the primary outcome being daily steps measured with motion sensors. The study will involve 252 patients from four spinal clinics. Get Back promotes increased physical activity and accessible rehabilitation, contributing to better health for LSS patients.

DETAILED DESCRIPTION:
The Get Back rehabilitation program has been developed using the Medical Research Councils (MRC) framework. A feasibility study (NCT05806593) has been completed involving 29 patients (mean age 67) who underwent surgery for LSS. The Get Back intervention (completely digital i.e. assessments and rehabilitation) was shown to be feasible and resulted in clinically significant improvements in daily steps at 12 weeks' post-surgery.

To evaluate the effectiveness and process of Get Back a multicenter randomized controlled trial including three sub-studies will be conducted. The specific research questions we aim to investigate in this RCT are:

1. if Get Back is more effective than standard rehabilitation in increasing daily steps (primary outcome) and physical activity behavior, disability, or pain-related factors (secondary outcomes) after surgery for LSS
2. if Get Back is more cost effective than standard rehabilitation after surgery for LSS
3. how baseline values (psychological factors, physical capacity and physical activity) predict changes in daily steps after surgery for LSS
4. how participants' experiences contribute to an enhanced understanding of what impact the intervention content had on their physical activity behavior.

Patients will be recruited from four clinical study sites (two private spine clinics and two hospitals). All patients undergo a clinical examination by an orthopedic surgeon as part of standard preoperative care. If a surgical decision is made and the patient is placed on the waiting list, a local recruiter at each site will hand out written study information to the patients meeting inclusion criteria and ask if a physical therapist from the study can make contact to provide further information about the study and ask for participation. As the intervention is fully digital, the patient information in written will also be sent to the patient digitally.

At baseline (approx. 2 weeks pre-surgery), participants meet with an assessor (physical therapist) via a digital care platform for collection of demographic data, personal goals, and to conduct physical capacity tests. Questionnaires are sent out through a digital application and patients wear an accelerometer for 7 days sent out by mail. Outcome variables are described more in detail under the heading Outcome Measures in the trial registration. The follow-ups are scheduled at 6 weeks, 3 months, 6 months, and 1-year post-surgery. Accelerometry and questionnaires will be collected at each follow-up, whereas physical capacity tests will be conducted at 3 and 12 months post-surgery. Clinical data such as type of surgery, complications, discharge destination will be collected from the patients' medical records at 3 months post-surgery.

After baseline assessments, patients are randomly assigned (1:1) to either control or intervention group. The randomization will be based on a computerized random list converted to concealed envelopes. The assessor will be blinded to group allocation.

Participants in the intervention group (Get Back, n=126) will have one pre-surgery video session with a physical therapist, followed by up to five core video sessions and five booster telephone sessions over 13 weeks. Session frequency is decided collaboratively, based on person-centered care. The intervention includes three components: graded physical activity, addressing fear avoidance beliefs, and promoting behavior change. A person-centered health plan is created at the first session, based on the patient's story and baseline assessment. The plan includes personalized activity goals, monitored using a weekly physical activity diary to track steps, barriers, and progress. A sub-sample of the intervention group, approximately 15-20 participants, will be interviewed regarding their experiences of the intervention and intervention content at 3 months post-surgery using a semi-structured interview guide.

Participants in the control group (n=126) will follow standard rehabilitation (physical therapy as provided at each site). Data on the frequency and content of rehabilitating sessions during the study will be collected as a control variable at each follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for decompression surgery due to central lumbar spinal stenosis

Exclusion Criteria:

* Patients with malignancy under treatment or with metastases;
* History of neurological or other disorders resulting in severe movement dysfunction;
* Untreated or instable heart conditions that prohibits physical tests;
* Poor understanding of Swedish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Steps per day collected with a activity tracker/accelerometer (Actigraph GT3X+). | At preoperative baseline, and at 6 weeks, 3 months, 6 months, 12 months postoperative follow-up
  Reported as number of steps per day. The primary endpoint is 3 months postoperatively.

SECONDARY OUTCOMES:
Physical activity level collected with a activity tracker/accelerometer (Actigraph GT3X+). | At preoperative baseline, and at 6 weeks, 3 months, 6 months, 12 months postoperative follow-up
  Reported as time spent in light physical activity, moderate to vigorous physical activity (MVPA) and time spent sedentary.
Physical function measured with the Timed-up-and-go test (TUG). | At preoperative baseline, 3 and 12 months postoperative follow-up.
  The time it takes for a participant to rise from a chair, walk 3 meters, turn, walk back to the chair and sit down. Reported in seconds.
Postural balance measured with the One Leg Stand test. | At preoperative baseline, 3 and 12 months postoperative follow-up.
  The time a participant can stand on one leg, reported in seconds.
Functional leg strength measured with the 30 seconds sit-to-stand test. | At preoperative baseline, 3 and 12 months postoperative follow-up.
  Reported as the number of chair rises a participant can complete during 30 seconds.
Pain intensity level in the leg and back reported with the Numeric Rating Scale (NRS). | At preoperative baseline, and at 6 weeks, 3 months, 6 months, 12 months postoperative follow-up.
  On a scale from 0 to 10, where a higher reported number means higher pain intensity.
Self-reported back-related disability collected with the Oswestry Disability Index (ODI). | At preoperative baseline, 3 and 12 months postoperative follow-up.
  Score range from 0 to 50. Higher scores represent greater disability.
The person's own goals regarding function collected with the Patient Specific Functional Scale (PSFS). | At preoperative baseline, 3 and 12 months postoperative follow-up.
  The participant will choose three activities of individual importance and rate the ability to perform each activity on a scale from 0 (not able to perform the activity) to 10 (can perform the activity unhindered).
Catastrophizing thoughts related to pain collected with the Pain Catastrophizing Scale (PCS). | At preoperative baseline, and at 6 weeks, 3 months, 6 months, 12 months postoperative follow-up
  Score range from 0 to 52. Higher scores mean higher degree of catastrophizing thoughts related to pain.
Patient-reported kinesiophobia collected with the Swedish version of the Tampa Scale of Kinesiophobia (TSK-SV). | At preoperative baseline, and at 6 weeks, 3 months, 6 months, 12 months postoperative follow-up.
  Score range from 17 to 68. Higher scores mean higher degree of fear of movement.
Depressed mood collected with the depression subscale of the Hospital Anxiety and Depression Scale. | At preoperative baseline, and at 6 weeks, 3 months, 6 months, 12 months postoperative follow-up.
  Score range from 0 to 21. A score of 8 or more indicates depression.
Pain self-efficacy collected with the 2-item Pain Self-Efficacy Questionnaire (PSEQ-2). | At preoperative baseline, and at 6 weeks, 3 months, 6 months, 12 months postoperative follow-up.
  The questions are rated on a scale from 0 (not at all confident) to 6 (completely confident). A score of 5 or less indicates that the person might be in need of help with their confidence in functioning in the presence of their pain. A score of 8 or higher reflects a desirable level of pain self-efficacy or confidence in functioning in the presence of pain.

OTHER OUTCOMES:
Direct costs, indirect costs and productivity losses collected with a self-report questionnaire. | At 6 weeks, 3, 6 and 12 months postoperative follow-up.
  Data for the health economic evaluation. A questionnaire including 10 questions (as well as subsections) aiming to capture costs from a societal perspective including direct costs (consultations, medical use, hospital stays), indirect (transportation), and productivity losses (sick leave) based on participants self-report. Treatment adherence and trial treatment costs, including education, the digital platform, and intervention materials, will be collected by the study physical therapist.
Health related quality of life collected with the EuroQol five dimension scale (EQ-5D 3L) | At preoperative baseline, and at 6 weeks, 3 months, 6 months, 12 months postoperative follow-up.
  Data for the health economic evaluation. Reported as an index utility score between 0 to 1 (a higher score indicates better health state) and a visual analogue scale of self-related overall health ranging from 0 to 100 (a higher score indicates better overall health).
Participants experiences of the intervention content collected via telephone interviews. | At 3 month postoperative follow-up (post-intervention).
  Semi structured telephone interviews with participants from the intervention group, which will be audio recorded and transcribed into text material.
Patient perceptions of person-centered care rated with the Generic Person-Centered Care Questionnaire (GPCCQ). | At 3 months postoperative follow-up.
  The questionnaire involves 18 questions answered on a 5-point scale where 1 ="No, not at all", and 5="Yes, completely". A higher scores mean a higher perception of person-centered care being present in the care.

CONTACTS AND LOCATIONS:
Overall Officials: Mari K Lundberg, Principal Investigator — Sophiahemmet University/Sophiahemmet Högskola
Locations (4):
- Sweden (4):
  - Ryggkirurgiskt centrum Stockholm, Stockholm
  - Södersjukhuset, Stockholm
  - Akademiska sjukhuset, Uppsala
  - Capio Spine Center Göteborg, Västra Frölunda

IPD SHARING:
Plan to Share IPD: No
The data in the study will be pseudonymized (coded) personal data, and Swedish legislation prohibits us from sharing this completely open. Some data is available upon request, which will be handled according to the relevant legislation.